CLINICAL TRIAL: NCT06027554
Title: The Mito-Frail Trial: Effects of MitoQ on Vasodilation, Mobility and Cognitive Performance in Frail Older Adults
Acronym: Mito-Frail
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Connecticut (Other)
Responsible Party: Principal Investigator, Oh Sung Kwon, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-132S-1; 1K01AG080164-01 (NIH); AG220138 (Other Grant/Funding Number: Patterson Trust)
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-01

CONDITIONS: Frailty; Mild Cognitive Impairment; Aging
MeSH Terms: conditions — Frailty; Cognitive Dysfunction | interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo capsule (Placebo Comparator): Gelatin capsules
  Interventions: Dietary Supplement: Placebo capsule
- MitoQ capsule (Experimental): Capsules containing mitoquinone mesylate (MitoQ, 5 mg/capsule) totaling 20 mg taken every day for 12 weeks.
  Interventions: Drug: Mitoquinone Mesylate

INTERVENTIONS:
Drug: Mitoquinone Mesylate — MitoQ given 20 mg per day for 12 weeks.
  Arms: MitoQ capsule
Dietary Supplement: Placebo capsule — Placebo capsule taken every day for 12 weeks.
  Arms: Placebo capsule

SUMMARY:
The goal of this clinical trial is to test the effects of MitoQ supplementation in older adults and frail older adults with physical dysfunction and/or cognitive dysfunction. The main question[s] it aims to answer are:

* To compare vascular function, oxidative stress levels, and physical and cognitive function among older adults and frail older adults with physical and cognitive dysfunction
* To determine whether MitoQ supplementation has the potential to improve vascular function in central and cerebral vessels
* To determine whether MitoQ supplementation can enhance physical and cognitive capabilities.

DETAILED DESCRIPTION:
Chronic diseases and associated declines in physical and cognitive performance contribute greatly to lost independence with aging. In addition to a lack of effective interventions other than exercise to address either problem, few studies have examined strategies for targeting both conditions in frail individuals who may experience difficulties with both walking and memory. Use of geroscience-guided therapies permits us to target mechanisms shared by aging with chronic conditions for which aging represents a major risk factor. Thus, instead of focusing on one single disease at a time, it may be possible to delay the onset and progression of disability involving multiple functional domains.

Gait speed is predictive of mobility, morbidity, and mortality in older adults. Vasoreactivity is a critical cerebrovascular control mechanism used to maintain brain perfusion during metabolic demands such as walking. In contrast to healthy older adults, middle cerebral artery blood flow velocities fail to increase proportionally in response to walking speed in slow walkers. Thus, abnormalities in vasoreactivity and perfusion adaptation to metabolic demands may reflect and contribute to declines in gait speed.

Mild cognitive impairment (MCI), an intermediate condition between normal cognitive performance and dementia, significantly increases the risk of transitioning dementia caused by Alzheimer's disease (AD). Moreover, changes in physical and cognitive function frequently co-exist in the same individual and influence each other.

In the absence of other effective therapies, modifiable cardiovascular risk factors (e.g., hypertension, atherosclerosis, cerebral hypoperfusion) represent opportunities to prevent declines in physical and cognitive function by targeting the vascular endothelium and vasodilation.

Physiological reactive oxygen species (ROS) levels play critical roles in cerebral vasculature, which can contribute to the regulation of brain perfusion through their action in vascular tone control. Of the many potential cellular sources of ROS in the vasculature, mitochondria are the major source in endothelium regulation of vascular homeostasis and are associated with aging and cardiovascular disease. Specifically, mitochondrialtargeted antioxidant, MitoQ, improves vascular endothelial function by reducing mitochondrial ROS (mtROS) in older adults and animal models.

Investigators have recently shown that MitoQ, a mitochondria-targeted antioxidant known to improve endothelial function and Nitric Oxide (NO) bioavailability, also restore impaired flow-mediated vasodilation in frail older adults, enhancing gait speed. In the Mito-Frail study, investigators will explore the hypothesis that MitoQ attenuates aging-related declines in flow-mediated vasodilation involving both peripheral and cerebral blood vessels. At the same time, investigators will obtain feasibility and pilot data involving measures of physical mobility and cognitive performance that may help us design and power a future clinical trial. Thus, this study will seek to develop strategies for preventing or slowing the progression of Alzheimer's Disease and the vascular contribution to dementia.

Therefore, Aim 1 will assess peripheral and cerebral NO bioavailability and mitochondrial reactive oxygen species (mtROS) levels in older adults who are healthy, others who are frail with slow walking speed and those who meet criteria for mild cognitive impairment (MCI). Aim 2 will determine whether MitoQ supplementation can enhance NO bioavailability and improve declines in flow-mediated vasodilation central and cerebral vessels.

Moreover, this study will also generate physical performance and cognitive data needed to design and power a future clinical trial focused on these functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 65-80 with a slow gait speed (0.4m/s based on a 4m walk) and/or mild cognitive impairment.
* good cardiovascular health (not taking any blood pressure/flow/metabolism altering medications)

Exclusion Criteria:

* A vaccination in past two weeks
* Recent acute infection three weeks prior to enrollment
* Known immunodeficiency (including HIV infection, primary immunodeficiency, any history of chemotherapy or radiotherapy
* Use of medicines during past 6 months known to alter immune response such as high- dose corticosteroids
* Severe autoimmune disease requiring biological therapy
* Major severe illness and/or Hospitalization in past 3 months
* On warfarin or other medications that are considered a blood thinner
* Recent fall or other conditions that will impair ability to complete and/or interpret mobility performance test
* Known bleeding disorder
* Any conditions that would impair the function to perform grip strength test
* include advanced neurological disease, severe co-morbid disease, terminal illness with reduced life expectancy, severe disability, unintentional weight loss in last 12 months and participation in another study.
* Diabetes patients requiring insulin (For reducing the risk that participants will have hypoglycemic episodes when fasting for study visits)
* Baseline ECG QTc >450 ms in men and QTc >460 ms in women
* Prior diagnosis of ventricular arrhythmia (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Vascular Endothelial Function | 4 visits : Baseline, 12 weeks (MitoQ or Placebo), 8 weeks washout, 12 weeks (MitoQ or Placebo)
  Assess Femoral artery through Passive Leg Movement and Brachial artery flow-mediated dilation (% [relative] and mm [absolute])
Change in Cerebrovascular Function | 4 visits : Baseline, 12 weeks (MitoQ or Placebo), 8 weeks washout, 12 weeks (MitoQ or Placebo)
  Utilize ultrasound to measure a change in blood flow velocity in response to a breathing test (cm/s)
Change in NIH Tool Box Composite | 4 visits : Baseline, 12 weeks (MitoQ or Placebo), 8 weeks washout, 12 weeks (MitoQ or Placebo)
  NIH Toolbox Cognitive Battery is a multidimensional set of brief measures assessing cognitive (as well as emotional, motor and sensory) function. There is no score range, but mean score is 100 with standard deviation 15. A score at or near 100 indicates average ability compared with others. Scores around 115 suggest above-average ability. Scores around 130 suggest superior ability (in the top 2 percent nationally). A score around 85 suggests below-average ability. A score in the range of 70 or below suggests significant impairment.
Change in walking speed | 4 visits : Baseline, 12 weeks (MitoQ or Placebo), 8 weeks washout, 12 weeks (MitoQ or Placebo)
  Gait speed calculated from 10 meter walk test. Only the 6 intermediate meters are recorded. Time is recorded by a manual chronometer. 3 records are done, mean time is calculated. Mean time is divided by 6 to obtain mean gait speed
Sensitivity of a Montreal Cognitive Assessment score | 4 visits : Baseline, 12 weeks (MitoQ or Placebo), 8 weeks washout, 12 weeks (MitoQ or Placebo)
  sensitivity of a Montreal Cognitive Assessment score < 26 to detect cognitive impairment defined as an abnormal result in at least one of the following tests : Test of Attentional Performance of Zimmermann and and Fimm (< 5th percentile in at least one of the subscales) ; Wechsler Adult Intelligence Scale 4th version digit span (standard score ≤ 5) ; Wechsler memory scale III, spatial span (standard score ≤ 5) ; Wisconsin Card Scoring Test, GREFEX version (number of categories ≤ 5th percentile or if the number of perseverations is ≥ 95th percentile) Wechsler Adult Intelligence Scale 4th version block design (standard score ≤ 5) ; Six elements test GREFEX version (rank score ≤ 5th percentile ); free and cued selective reminding test, 16 items, B version (Z-score ≤ -1,65 in at least one of the subscales)

SECONDARY OUTCOMES:
Change in Mitochondrial Function measured in peripheral blood mononuclear cells (PBMCs) | 4 visits : Baseline, 12 weeks (MitoQ or Placebo), 8 weeks washout, 12 weeks (MitoQ or Placebo)
  Measure mitochondrial respiratory function using peripheral blood mononuclear cells (PBMCs) using oroboros O2k system expressed by O2flux in pmol/second/cell numbers
Change in Oxidative Stress measured in peripheral blood mononuclear cells (PBMCs) by O2flux in pmol/second/cell numbers | 4 visits : Baseline, 12 weeks (MitoQ or Placebo), 8 weeks washout, 12 weeks (MitoQ or Placebo)
  Measure Mitochondrial-derived reactive oxygen species (ROS) using peripheral blood mononuclear cells (PBMCs) using oroboros O2k system expressed by Amplex flux in pmol/second/cell numbers

CONTACTS AND LOCATIONS:
Overall Officials: Oh Sung Kwon, PhD, Principal Investigator — University of Connecticut
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No